CLINICAL TRIAL: NCT04241029
Title: Boosting Biologics in Ulcerative Colitis
Brief Title: Boosting Biologics in UC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: Helse Sor-Ost (Other Government)
Responsible Party: Principal Investigator, Asle W. Medhus, Head of dep. of Gastroenterology, OUH. MD, PhD., Oslo University Hospital
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2016/2269
Record Dates: First submitted 2020-01-17; First posted 2020-01-27 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: Ulcerative Colitis; Inflammatory Bowel Diseases
MeSH Terms: conditions — Colitis, Ulcerative; Inflammatory Bowel Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention with probiotics (Experimental): Intervention with the probiotic compound IDOFORM®Travel. The patient will receive four capsules orally every 24 hour (12*10^9 cfu/day) for eight weeks as adjuvant therapy to his/her anti-TNF treatment. The intervention arm will at the end of intervention serve as their own controls compared to baseline data (before intervention).
  Interventions: Dietary Supplement: IDOFORM®Travel

INTERVENTIONS:
Dietary Supplement: IDOFORM®Travel — Four capsules IDOFORM®Travel orally every 24 hour (12*10^9 cfu/day) for eight weeks.

SUMMARY:
This study evaluates the safety of the probiotic compound IDOFORM TRAVEL® in patients with ulcerative colitis undergoing anti-TNF treatment with insufficient clinical response. Furthermore, the study aims to explore the composition of the bacteria of the gut as well as the immunological activity in patients with ulcerative colitis undergoing anti-TNF treatment, aiming to identify differences between groups of patients responding and not responding adequately to treatment.

The project will explore whether probiotics have beneficial effects as adjuvant therapy in ulcerative colitis patients with insufficient response to anti-TNF treatment.

DETAILED DESCRIPTION:
The use of anti TNF agents has improved the medical treatment of ulcerative colitis (UC). However, one third of patients receiving such treatment will not reach remission. Studies have demonstrated that the gut microbiome influences the cytokine response and in particular the TNF production. In this study we aim to manipulate the gut microbiome in patients with ulcerative colitis not responding to anti-TNF therapy to evaluate potential beneficial effects.

20 UC patients with insufficient response to anti-tumor necrosis factor (anti-TNF) therapy upon routine evaluation colonoscopy 6-12 months after start of treatment will receive intervention with the probiotic formula IDOFORM Travel®, 4 capsules daily for 8 weeks. A colonoscopy will be performed at baseline (week 0) and after intervention (week8). Gut biopsies, fecal samples and serological markers will, in addition to clinical examination and endoscopic results, be used to evaluate the safety and possible beneficial effects of the intervention.

In a subsidiary cross-sectional study, 20 UC patients on anti-TNF therapy in remission upon evaluation colonoscopy will serve as controls. 20 individuals with no history of inflammatory bowel disease will be recruited as healthy controls.

ELIGIBILITY:
Inclusion Criteria:

Subjects may be included as cases in the study if they meet all of the following criteria:

* Diagnosed With ulcerative colitis based on Lennard-Jones criteria
* Under treatment With anti-TNF infusions/injections defined as infliximab or adalimumab
* Failure to Reach remission upon routine evaluation colonoscopy after 6-12 months of treatment - defined as an endoscopy sub score of ≥ using the Mayo score for ulcerative colitis
* Age 18-75
* Signed informed consent and expected Cooperation of the patients for the treatment and follow up must be obtained and documented according to International Committee on Harmonization (ICH) Good Clinical Practice (GCP), and national/local regulations.

Subjects may be included as Control subjects in the sub-study if they meet all of the following criteria:

* Diagnosed With ulcerative colitis based on Lennard-Jones Criteria
* Under treatment With anti-TNF infusions/injections defined as infliximab or adalimumab
* Remission upon routine colonoscopy after 6-12 months of treatment - defined as an endoscopy sub score of ≤ using the Mayo score for ulcerative colitis
* Age 18-75
* Signed informed consent and expected Cooperation of the patients for the treatment and follow up must be obtained and documented according to International Committee on Harmonization (ICH) Good Clinical Practice (GCP), and national/local regulations.

OR if they meet all the following criteria:

* No history of inflammatory bowel disease
* Age 18-75
* Signed informed consent and expected Cooperation of the patients for the treatment and follow up must be obtained and documented according to International Committee on Harmonization (ICH) Good Clinical Practice (GCP), and national/local regulations.

Exclusion Criteria:

* Clinical status poor to such extent that treating physician finds refraining from escalation of treatment contraindicated
* Signs of severe ulcerative colitis as defined by the "Montreal classification of severity of ulcerative colitis" = 3: Passage of at least six bloody stools daily, pulse rate of at least 90 beats per minute, temperature of at least 37.5°C, haemoglobin of less than 10.5 g/100 ml, and erythrocyte sedimentation rate (ESR) of at least 30 mm/h.
* Previous use of anti-TNF medication
* History of bowel resection, other inflammatory bowel disease (IBD)-related surgery, or other major intestinal surgery
* Plasma hepatitis C (HCV) positive
* Serum hepatitis B surface antigen (HBsAg) positive
* HIV positive
* Comorbidity of coeliac disease or malnutrition
* Pregnancy
* Concomitant use of non-steroid anti-inflammatory drugs (NSAIDS) or corticosteroids
* Concomitant use of antithrombotic pharmaceutical substances
* Regular (weekly) use of any probiotic substance within 3 months prior to inclusion
* Use of antibiotics within 3 months prior to inclusion
* Deranged liver function (serum albumin < 25 g/L or Child-Pugh ≥10)
* Renal failure (estimated glomerular filtration rate (eGFR) < 30
* Heart failure (NYHA class II-IV)
* Any reason why, in the opinion of the investigator, the patient should not participate

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2020-02-25 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
Adverse events | 8 weeks
  Unit of Measure: Frequency
Total Mayo Score for Ulcerative Colitis | 8 weeks
  Alterations in Total Mayo Score at time of control colonoscopy. Minimal value=0 (best outcome), Maximal value = 12 (worst outcome)
Change in Fecal Calprotectin | 12 weeks
  Change in Fecal Calprotectin from baseline (week 0) to end of intervention (week 8) and after intervention (week 12).
  Unit of measure: mg/kg

SECONDARY OUTCOMES:
Alterations in mucosa-adherent microbial composition | 8 weeks
  Exploratory analyses of microbial composition at baseline (week 0) and at end of intervention (week 8). (Unit of Measure: Descriptive)
Alterations in epithelial gene expression | 8 weeks
  Exploratory (Unit of Measure: Descriptive)
Alterations in markers of chronic inflammation / immune activation | 8 weeks
  Explorative (Unit of Measure: Descriptive)

CONTACTS AND LOCATIONS:
Overall Officials: Asle Medhus, MD, PhD, Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Oslo, Norway